CLINICAL TRIAL: NCT03444012
Title: Non-interventional Prospective Data Collection on Persistence and Adherence on Ticagrelor in ACS Adult Patients in Serbia
Brief Title: ADHERE-S (NIS Brilique)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5130R00052
Record Dates: First submitted 2018-02-09; First posted 2018-02-23 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: ACS (Acute Coronary Syndrome)
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

INTERVENTIONS:
Drug: ticagrelor 90 mg — persistence and adherence on ticagrelor in ACS patients

SUMMARY:
noninterventional study investigating persistence and adherence on ticagrelor in ACS patients in Serbia

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* diagnosed with ACS - STEMI or NSTEMI or unstable angina, invasively or non-invasively treated
* Patients already on treatment with ticagrelor at least for 1 month and no longer than 3 months prior to study initiation. Enrolment in this study must not be trigger for ticagrelor initiation.
* read and signed the Informed Consent Form

Exclusion Criteria:

Any contraindications as per approved SmPC of Brilique

• Patients with life-threatening conditions which could disable patients to comply with scheduled visits and/or not able to fill in the patient questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ACS patients
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
duration (number of days) on ticagrelor therapy in patients with acute coronary syndrome | 1 year (12 months)

CONTACTS AND LOCATIONS:
Locations (9):
- Serbia (9):
  - CHC Bezanijska Kosa, Belgrade
  - CHC Zemun, Belgrade
  - CHC Zvezdara, Belgrade
  - Clinical Center of Serbia, Belgrade
  - Institute for cardiovascular diseases, Dedinje, Belgrade
  - Medical Military Academy, Belgrade
  - Institute for cardiovascular diseases of Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš

REFERENCES:
- See also: redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5130R00052&attachmentIdentifier=fbea9a76-9c50-468b-853b-dc84feb338df&fileName=D5130R00052_CSR_Synopsis.pdf&versionIdentifier=